CLINICAL TRIAL: NCT01648621
Title: Program of Integrated Care for Patients With Chronic Obstructive Pulmonary Disease and Multiple Comorbidities: A Randomized Controlled Trial
Brief Title: Program of Integrated Care for Patients With Chronic Obstructive Pulmonary Disease and Multiple Comorbidities
Acronym: PICCOPD+
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michael Garron Hospital (Other)
Collaborators: Southlake Regional Health Centre (Other); University of Toronto (Other); Ontario Ministry of Health and Long Term Care (Other Government)
Responsible Party: Principal Investigator, Louise Rose, Director of Research, Prolonged ventilation Weaning Centre, Michael Garron Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TEGH001 PIC COPD
Record Dates: First submitted 2012-07-19; First posted 2012-07-24 (Estimated); Last update posted 2016-11-11 (Estimated); Status verified 2016-11

CONDITIONS: Chronic Obstructive Pulmonary Disease; Multiple Comorbidity
Keywords: COPD; case management
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Case Management (Experimental): In addition to usual care, the intervention group will receive case management that includes: 40 minute standardized education session, an individualized action plan, an individualized care plan for management of COPD and comorbidities, standardized reinforcement/motivational interviewing and action plan teach-back sessions and assessment of symptoms, progress and problems, and problem solving by phone weekly for 12 weeks, then monthly for 9 months (21 sessions), tele-home monitoring, coordinated and improved communication between the patient, family caregivers, family physicians, specialists, and CCAC facilitated by the case manager, priority access to ambulatory clinics.
  Interventions: Behavioral: 40 minute standardized education session; Behavioral: Individualized action plan; Behavioral: Individualized care plan; Behavioral: Standardized reinforcement/motivational interviewing and action plan teach-back sessions; Behavioral: Tele-home monitoring; Behavioral: Coordinated and improved communication; Behavioral: Priority access; Behavioral: Dictated patient summary; Behavioral: in-hospital rehabilitation/self-management program; Behavioral: Smoking cessation
- Usual care (Active Comparator): Usual care for these patients comprises: Dictated patient summary, referral to an 8 week in-hospital rehabilitation and self-management education program, referral to a smoking cessation program (as applicable), individualized action plan developed with treating respirologist at the discretion of the attending respirologist, Referral to web based educational materials and resources.
  Interventions: Behavioral: Dictated patient summary; Behavioral: in-hospital rehabilitation/self-management program; Behavioral: Smoking cessation; Behavioral: Action plan Respirologist; Behavioral: Web based self management materials

INTERVENTIONS:
Behavioral: 40 minute standardized education session — 40 minute standardized education session based on the Living Well with COPD Patient's Education Tool on study enrolment to assess and improve understanding of disease and ability to monitor symptoms and recognize exacerbation
  Arms: Case Management
Behavioral: Individualized action plan — Individualized action plan using the Living Well with COPD template with patient individualized modification to address management strategies for exacerbation of comorbidity developed during the initial 40 minute session with case manager.
  Arms: Case Management
Behavioral: Individualized care plan — Individualized care plan for management of COPD and comorbidities developed by the case manager in consultation with family physician and specialists.
  Arms: Case Management
Behavioral: Standardized reinforcement/motivational interviewing and action plan teach-back sessions — Standardized reinforcement/motivational interviewing and action plan teach-back sessions based on Living Well with COPD modules as well as assessment of symptoms, progress and problems, and problem solving by phone weekly for 12 weeks, then monthly for 9 months (21 sessions) (telephone script; NOTE: case managers will make up to 3 attempts to contact participants during each week of the 12 weeks of weekly phone calls before determining inability to contact the participant for that week.
  Arms: Case Management
Behavioral: Tele-home monitoring — Tele-home monitoring of SpO2, weight, dyspnea, sputum quantity and characteristics, and general well-being for maximum of 6 months.
  Inclusion criteria for tele-home monitoring:
  a. compatible phone line b. patient consent c. patient or caregiver demonstrated ability to use monitoring equipment d. patient unable to attend outpatient/community appointments for assessment and monitoring because of environmental barriers to access (e.g. physician's office only accessible by stairs) e. severe dyspnea on activities of daily living (Medical Research Council Questionnaire for Assessing Severity of Breathlessness [MRC] Class 4 & 5 or modified MRC [mMRC] 3 & 4) f. frequent ED visits (> 2) in last 12 months
  5. 12 weeks of clinical stability with no ED visits.
  Arms: Case Management
Behavioral: Coordinated and improved communication — Coordinated and improved communication between the patient, family caregivers, family physicians, specialists, and Community Care Access Centres (CCACs) facilitated by the case manager. This will include phone contact by case manager to family physicians and CCAC case manager if applicable after initial enrollment, education session and development of action plan, then monthly to report general status as well as after subsequent ED presentations/hospital admissions
  Arms: Case Management
Behavioral: Priority access — Priority access to ambulatory clinics (Respirology and other specialties as required including Psychiatry) facilitated through the case manager.
  Arms: Case Management
Behavioral: Dictated patient summary — Dictated patient summary sent by specialists (e.g. respirologists) to family physicians following each respiratory centre visit (every 12 weeks)
Behavioral: in-hospital rehabilitation/self-management program — Referral to an 8 week in-hospital rehabilitation and self-management education program for patients that are:
  1. have had a recent exacerbation, but are now clinically stable;
  2. symptomatic COPD including reduced activity levels and increased dyspnea despite pharmacological treatment;
  3. have stabilized comorbidity (no evidence of active ischemic, musculoskeletal, psychiatric or other systemic disease); and
  4. have sufficient motivation to participate.
Behavioral: Smoking cessation — Referral to a smoking cessation program (as applicable)
Behavioral: Action plan Respirologist — Individualized action plan developed with treating respirologist at the discretion of the attending respirologist.
  Arms: Usual care
Behavioral: Web based self management materials — Referral to educational materials and resources (Living Well with COPD module printouts provided during COPD rehabilitation classes at a cost to the individual)
  Arms: Usual care

SUMMARY:
Many patients with chronic obstructive pulmonary disease (COPD) also have other diseases referred to as comorbidities. Often these patients require health care by a variety of health care professionals from services linked to hospitals and in the community. Unfortunately, sometimes it may be difficult for these patients to receive appropriate care in a timely manner resulting in a trip to the emergency department. As well, patients may benefit from education that enables them to recognize early signs indicating they are getting sicker and to self-manage their disease. Our study will examine a strategy that includes a case manager who will make weekly phone contact with COPD patients with comorbidity that present either to the emergency department or are admitted to hospital. Weekly contact will focus on teaching patients to recognize worsening symptoms and self-management strategies. The case manager will work with patients, caregivers, community health care providers and hospital specialists to promote communication and optimize care delivery. The investigators will examine the impact of our intervention on the need for emergency department visits and hospital admission. The investigators will also examine the impact on patients' health related quality of life, number of COPD exacerbations, and disease progression.

ELIGIBILITY:
Inclusion Criteria:

* COPD defined as chronic irreversible airflow limitation with FEV1 < lower limit of normal for age as % predicted and a FEV1/FVC ratio < than lower limit of normal (usually 70%) [5]

Plus ≥ 2 comorbidities commonly associated with COPD as identified in the Canadian Thoracic Society COPD guidelines*

1. Cardiovascular disease
2. Osteopenia and osteoporosis
3. Glaucoma and cataracts
4. Cachexia and malnutrition
5. Peripheral muscle dysfunction
6. Lung cancer
7. Metabolic syndrome (diabetes mellitus)
8. Depression
9. Chronic kidney disease OR Other conditions as primary admitting/presenting diagnosis + COPD as significant comorbidity + ≥ 1 other comorbidity

THAT

1. Get admitted to participating hospital; or
2. Present to participating hospital ED; or
3. Have first referral to Respiratory Centre/Respirology team

AND HAVE

1. ≥ 1 ED presentation/hospital admission in previous 12 months
2. ≥ 50 years age

Exclusion Criteria:

1. No access to primary care physician
2. Primary diagnosis of asthma
3. Terminal diagnosis (metastatic disease with a life expectancy of ≤ 6 months)
4. Dementia and absence of family caregiver able to assist with activation of the action plan and feedback on ongoing status and care coordination
5. Uncontrolled psychiatric illness
6. Inability to understand, read, and write English
7. No access to a phone
8. Inability to attend follow up at one of the participating sites

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 470 (Actual)
Dates: Start 2012-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
The number of ED presentations | 1 year after randomization.

SECONDARY OUTCOMES:
Hospital admission rates | 1 year after randomization
Number of hospitalized days over 1 year | At one year after randomization
Time to death | During 12 months of intervention
COPD severity measured by the BODE index | at baseline, 6 months and 1 year
  The BODE Index is a simple grading system for COPD comprising the Six Minute Walk Distance (6MWD), the Medical Research Council Dyspnea Scale (MMRC) and body mass index (BMI).
Change in health-related quality of life | baseline at 90 days, 6 months and 1 year
  Measured using the EQ5D, St George's Respiratory Questionnaire, Hospital Anxiety and Depression Scale (HADS)
Change in COPD self-efficacy scale | baseline at 90 days, 6 months and 1 year
  The COPD SES provides items with sufficient complexity in relation to the specific situation of managing with COPD. The CSES consists of Likert scale with 5 responses from "very confident" to "not at all confident" scoring 5 to 1 with 5 representing higher self-efficacy.
Patient satisfaction using the CSQ8 | 90 days, 6 months and 1 year
Caregiver impact (Caregiver Impact Scale) | at baseline, 6 months and 1 year
  This questionnaire assesses the impact of caregiving on 14 different domains (health, employment, family relations), using a 7-point Likert scale.

OTHER OUTCOMES:
Adherence to chronic disease management measures | at 1 year
  smoking cessation status (if applicable), influenza and pneumonia vaccination, up-to-date documented action plan, electronic medication reconciliation

CONTACTS AND LOCATIONS:
Overall Officials: Louise Rose, PhD, Principal Investigator — Toronto East General Hospital/University of Toronto; Ian Fraser, MD, Principal Investigator — Michael Garron Hospital
Locations (2):
- Canada (2):
  - Southlake Regional Heath Centre, Newmarket, Ontario
  - Toronto East General Hospital, Toronto, Ontario

REFERENCES:
- [Derived] Poot CC, Meijer E, Kruis AL, Smidt N, Chavannes NH, Honkoop PJ. Integrated disease management interventions for patients with chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2021 Sep 8;9(9):CD009437. doi: 10.1002/14651858.CD009437.pub3. PMID 34495549
- [Derived] Rose L, Istanboulian L, Carriere L, Thomas A, Lee HB, Rezaie S, Shafai R, Fraser I. Program of Integrated Care for Patients with Chronic Obstructive Pulmonary Disease and Multiple Comorbidities (PIC COPD+): a randomised controlled trial. Eur Respir J. 2018 Jan 11;51(1):1701567. doi: 10.1183/13993003.01567-2017. Print 2018 Jan. PMID 29326330